CLINICAL TRIAL: NCT07143994
Title: Eccentric vs. Concentric Training: Accelerating Recovery in Elite Athletes With Grade II Hamstring Injury
Brief Title: EFFECT OF ECCENTRIC AND CONCENTRIC EXERCISE PROGRAMS For HAMSTRING GRADE INJURIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Feyza Sule BADILLI HANTAL, Asst.Prof, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hamstring eccentring
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hamstring Injuries
Keywords: grade 2 muscle injury; eccentric exercise; concantric exercise; balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric Exercise Program (Experimental): Elite athletes with grade II hamstring strain will undergo a structured rehabilitation protocol consisting of eccentric strengthening exercises. The program is designed to improve hamstring flexibility, strength, dynamic balance, and facilitate safe return to sport.
  Interventions: Other: eccentric exercise
- Concentric Exercise Intervention (Experimental): Elite athletes with grade II hamstring strain will undergo a structured rehabilitation protocol consisting of concentric strengthening exercises. The program is designed to enhance hamstring flexibility, muscle strength, dynamic balance, and assist in safe return to sport.
  Interventions: Other: concentric exercise

INTERVENTIONS:
Other: eccentric exercise — This study's interventions are distinguished by the specific application of eccentric and concentric exercise programs tailored for elite athletes with grade II hamstring strains.
  Arms: Eccentric Exercise Program
Other: concentric exercise — This study's interventions are distinguished by the specific application of eccentric and concentric exercise programs tailored for elite athletes with grade II hamstring strains.
  Arms: Concentric Exercise Intervention

SUMMARY:
Hamstring injuries are common and recurrent in both elite and recreational athletes, often leading to prolonged absence from sports. The aim of this study is to compare the effects of eccentric and concentric exercise programs on the recovery of elite athletes diagnosed with grade II hamstring strain. Pain, flexibility, muscle strength, balance, and return-to-sport duration will be evaluated to determine the impact of different exercise modalities. Dynamic balance assessment will also be performed before and after treatment. The two intervention groups will be compared using the Wilcoxon test, with p<0.01 considered statistically significant. This study is expected to provide evidence on which exercise program is more effective in facilitating return to sport and to contribute to improved rehabilitation strategies in future athletic injuries.

DETAILED DESCRIPTION:
amstring muscle strain is one of the most common injuries in elite sports, frequently leading to long rehabilitation periods and a high rate of recurrence. Although various treatment modalities have been studied, there is still no consensus on the most effective exercise approach for recovery and return to sport. This study investigates the effectiveness of two different rehabilitation strategies-eccentric exercise programs and concentric exercise programs-in elite athletes diagnosed with grade II hamstring strain.

The intervention will focus on structured exercise protocols applied over a defined treatment period. Outcomes to be assessed include pain intensity, hamstring flexibility, isometric and isotonic muscle strength, dynamic balance, and time to return to sport. Dynamic balance assessment is included as a novel parameter to better understand functional recovery after hamstring injury.

Statistical analysis will be performed using the Wilcoxon test for continuous variables, with p<0.01 considered significant. The results are expected to clarify which type of exercise program provides superior outcomes in terms of functional recovery and safe return to sport. This may help guide clinicians in designing more effective rehabilitation strategies for elite athletes and reduce the recurrence of hamstring injuries.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 ,who are elite athlete and contunie currently active sports life,and . Those with MRI findings showing hamstring grade II strain,who does not have any systemic or mental disease volunteerly participated in the study.

Exclusion Criteria:

* Participants who are having severe visual impairment and perception impairment, who has pain preventing to test,who has neurologic problems ans who has a history of injury for 6 months were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Time to Return to Sport | From baseline until return to sport, up to 12 weeks
  he duration (in days) from the start of the rehabilitation program until the athlete meets all return-to-play criteria, including complete pain relief, sufficient muscle strength, joint mobility, flexibility, running and gait analysis, physical fitness, balance, dynamic functional performance, lumbopelvic motor control, and subjective readiness reported by the athlete.

CONTACTS AND LOCATIONS:
Locations (1):
- HANTAL, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding the sharing of individual participant data (IPD) has not yet been made. Considerations regarding participant privacy, confidentiality, and the sensitive nature of the data will inform any future decisions on data sharing.